CLINICAL TRIAL: NCT03361540
Title: A Placebo-controlled, Single and Multiple Ascending Oral Dose Study in Non-elderly Healthy Japanese Male and Female Subjects
Brief Title: ASP8302 Single and Multiple Ascending Oral Dose Study in Non-elderly Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: 8302-CL-0101
Record Dates: First submitted 2017-11-14; First posted 2017-12-05 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2019-04

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Safety; ASP8302

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Single dose of ASP8302 dose-1 (Experimental): Subjects will receive a single dose of ASP8302.
  Interventions: Drug: ASP8302
- Single dose of ASP8302 dose-2 (Experimental): Subjects will receive a single dose of ASP8302.
  Interventions: Drug: ASP8302
- Single dose of ASP8302 dose-3 (Experimental): Subjects will receive a single dose of ASP8302.
  Interventions: Drug: ASP8302
- Single dose of ASP8302 dose-4 (Experimental): Subjects will receive a single dose of ASP8302.
  Interventions: Drug: ASP8302
- Single dose of Placebo (Placebo Comparator): Subjects will receive a single dose of Placebo.
  Interventions: Drug: Placebo
- Multiple dose of ASP8302 dose-5 (Experimental): Subjects will receive once daily dosing of ASP8302 for 14 consecutive days at the same dose level.
  Interventions: Drug: ASP8302
- Multiple dose of ASP8302 dose-6 (Experimental): Subjects will receive once daily dosing of ASP8302 for 14 consecutive days at the same dose level.
  Interventions: Drug: ASP8302
- Multiple dose of Placebo (Placebo Comparator): Subjects will receive once daily dosing of Placebo for 14 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP8302 — ASP8302 will be administered orally.
  Arms: Multiple dose of ASP8302 dose-5; Multiple dose of ASP8302 dose-6; Single dose of ASP8302 dose-1; Single dose of ASP8302 dose-2; Single dose of ASP8302 dose-3; Single dose of ASP8302 dose-4
Drug: Placebo — Placebo will be administered orally.
  Arms: Multiple dose of Placebo; Single dose of Placebo

SUMMARY:
The objective of this study is to evaluate the safety, tolerability and pharmacokinetic of single/multiple ascending oral doses of ASP8302 in non-elderly healthy Japanese male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight at screening: ≥ 50.0 kg and < 80.0 kg for male, ≥ 40.0 kg and < 70.0 kg for female.
* Body-mass index (BMI) at screening: ≥ 17.6 kg/m2 and < 26.4 kg/m2 [BMI = Body weight (kg) ÷ {Body height (m)2}].

Exclusion Criteria:

* Subjects who participated or are scheduled to participate in any clinical trials or post-marketing studies within 120 days before screening test or during the screening test to the hospital admission (Day -2).
* Subjects who conducted or is scheduled to conduct any of the blood donation or blood drawing in designated period before Day -2
* Subject who received or is scheduled to receive any medications within seven days before the hospital admission.
* Any deviation from any of the normal range of blood pressure, pulse rate, body temperature and standard 12-lead electrocardiogram at screening or on the day of hospital admission (Day -1).
* Subject who meets any of the criteria for laboratory tests at screening or on the day of hospital admission (Day -2).
* Any deviation from the normal range of routine 12-lead electrocardiogram at screening.
* Subjects with a complication or history of drug allergies.
* Subjects who developed upper gastrointestinal symptoms within seven days before the hospital admission.
* Subjects with a complication or history of hepatic disease.
* Subjects with a complication or history of cardiac disease.
* Subjects with a complication or history of respiratory disease except for history of asthma in childhood.
* Subjects with a complication or history of gastrointestinal disease except for a history of appendicitis.
* Subjects with a history of gastrointestinal resection except for appendicitis.
* Subjects with a complication or history of renal disease except for a history of calculus.
* Subjects with a complication or history of endocrine disease.
* Subjects with a complication or history of cerebrovascular disease.
* Subjects with a complication or history of malignant tumor.
* Subjects who received ASP8302 previously.
* Subjects who have a habit of excessive smoking or drinking alcohol.

Ages: 20 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Safety assessed by incidence of adverse events (AEs) | Up to Day 6 in single ascending dose (SAD) part Up to Day 19 in MAD part
  Adverse events will be coded using Medical Dictionary for Regulatory Activities (MedDRA).
Safety assessed by vital signs: Body temperature | Up to Day 6 in SAD part Up to Day 19 in multiple ascending dose (MAD) part
  To assess vital signs as a criteria of safety variables.
Safety assessed by vital signs: Blood pressure | Up to Day 6 in SAD part Up to Day 19 in MAD part
  To assess vital signs as a criteria of safety variables.
Safety assessed by vital signs: Pulse rate | Up to Day 6 in SAD part Up to Day 19 in MAD part
  To assess vital signs as a criteria of safety variables.
Number of participants with laboratory value abnormalities and/or AEs | Up to Day 6 in SAD part Up to Day 19 in MAD part
  Number of participants with potentially clinically significant laboratory values.
Safety assessed by cardiac troponin | Up to Day 6 in SAD part Up to Day 19 in MAD part
  To assess the cardiovascular system function as a criteria of safety variables.
Safety assessed by standard 12-lead electrocardiogram | Up to Day 6 in SAD part Up to Day 19 in MAD part
  To assess the cardiovascular system function as a criteria of safety variables.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) parameter for ASP8302: Maximum observed concentration (Cmax) in plasma | Up to 72 hr after dosing in SAD part Day 1 and Day 14 in MAD part
  To assess the PK of ASP8302 in SAD part and MAD part.
PK parameter for ASP8302: Time of the Maximum Concentration (tmax) in plasma | Up to 72 hr after dosing in SAD part Day 1 and Day 14 in MAD part
  To assess the PK of ASP8302 in SAD part and MAD part.
PK parameter for ASP8302: Area under the concentration-time curve (AUC) from the time of dosing to 24h after dosing (AUC24) in plasma | Up to 72 hr after dosing in SAD part Day 1 in MAD part
  To assess the PK of ASP8302 in SAD part and MAD part.
PK parameter for ASP8302: AUC from the Time of Dosing Extrapolated to Time Infinity (AUCinf) in plasma | Up to 72 hr after dosing in SAD part
  To assess the PK of ASP8302 in SAD part.
PK parameter for ASP8302: AUC from the Time of Dosing to the Start of the Next Dosing Interval (AUCtau) in plasma | Day 14 in MAD part
  To assess the PK of ASP8302 in MAD part.
PK parameter for ASP8302: Peak-Trough Ratio (PTR) in plasma | Day 14 in MAD part
  To assess the PK of ASP8302 in MAD part.
PK parameter for ASP8302: Accumulation Ratio for AUC (Rac(AUC)) in plasma | Day 14 in MAD part
  To assess the PK of ASP8302 in MAD part.
PK parameter for ASP8302: Accumulation Ratio for Cmax (Rac(Cmax)) in plasma | Day 14 in MAD part
  To assess the PK of ASP8302 in MAD part.
PK parameter for ASP8302: AUC from the Time of Dosing to the Last Measurable Concentration (AUClast) in plasma | Up to 72 hr after dosing in SAD part
  To assess the PK of ASP8302 in SAD part.
PK parameter for ASP8302: Time Point Prior to the Time Point Corresponding to the First Measurable (Non-zero) Concentration (tlag) in plasma | Up to 72 hr after dosing in SAD part Day 1 in MAD part
  To assess the PK of ASP8302 in SAD part and MAD part.
PK parameter for ASP8302: Terminal Elimination Half-life (t1/2) in plasma | Up to 72 hr after dosing in SAD part Day 14 in MAD part
  To assess the PK of ASP8302 in SAD part and MAD part.
PK parameter for ASP8302: Apparent Volume of Distribution during the Terminal Elimination Phase After Single Extra-Vascular Dosing (Vz/F) in plasma | Up to 72 hr after dosing in SAD part
  To assess the PK of ASP8302 in SAD part.
PK parameter for ASP8302: Apparent Total Systemic Clearance After Single or Multiple Extra-Vascular Dosing (CL/F) in plasma | Up to 72 hr after dosing in SAD part Day 14 in MAD part
  To assess the PK of ASP8302 in SAD part and MAD part.
PK parameter for ASP8302: Concentration Immediately Prior to Dosing at Multiple Dosing (Ctrough) in plasma | Up to Day 14 in MAD part
  To assess the PK of ASP8302 in MAD part.
PK parameter for ASP8302: Amount excreted into urine from the time of dosing to the 72 hours after dosing (Ae72) in urine | Up to 72 hr after dosing in SAD part
  To assess the PK of ASP8302 in SAD part.
PK parameter for ASP8302: Fraction excreted into urine from the time of dosing to the 72 hours after dosing (Ae72%) in urine | Up to 72 hr after dosing in SAD part
  To assess the PK of ASP8302 in SAD part.
PK parameter for ASP8302: Renal clearance (CLR) in urine | Up to 72 hr after dosing in SAD part Day 14 in MAD part
  To assess the PK of ASP8302 in SAD part and MAD part.
PK parameter for ASP8302: Amount excreted into urine over the time interval between consecutive dosing (Aetau) in urine | Day 14 in MAD part
  To assess the PK of ASP8302 in MAD part.
PK parameter for ASP8302: Fraction excreted into urine over the time interval between consecutive dosing (Aetau%) in urine | Day 14 in MAD part
  To assess the PK of ASP8302 in MAD part.
Pharmacodynamic (PD) parameter for ASP8302: Pupil diameter | Up to 24 hr after dosing in SAD part Up to Day 14 in MAD part
  To assess the PD of ASP8302 in SAD part and MAD part.
PD parameter for ASP8302: Salivary secretion | Up to 24 hr after dosing in SAD part Up to Day 14 in MAD part
  To assess the PD of ASP8302 in SAD part and MAD part.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Toshima City, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.